CLINICAL TRIAL: NCT07375849
Title: Application of Electrical Impedance Tomography in Evaluating Pulmonary Function Improvement After High Lateral Recumbent Position Therapy in ARDS Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2025-143
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 90-degree high lateral position group (Experimental): Place the patient in the 90-degree high lateral position.
  Interventions: Procedure: Place the patient in the 90-degree high lateral position.
- 30-degree low lateral position group (Experimental): Place the patient in the 30-degree low lateral position.
  Interventions: Procedure: Place the patient in the 30-degree low lateral position.
- 120-degree high lateral position group (Experimental): Place the patient in the 120-degree high lateral position.
  Interventions: Procedure: Place the patient in the 120-degree high lateral position.
- Prone position group (Active Comparator): Patients will be placed in the prone position, i.e., lying face down.
  Interventions: Procedure: Patients will be placed in the prone position, i.e., lying face down.

INTERVENTIONS:
Procedure: Place the patient in the 90-degree high lateral position. — For the 90° lateral recumbent position group, patients will be rotated between corresponding lateral recumbent positions on the left and right sides every 2 hours, spending 8 hours on each side for a total treatment duration of 16 hours. During each rotation, the nursing team will ensure the patient is safely transferred from one side to the other while maintaining the prescribed lateral angle. Wedge pillows or specialized turning pads will be used to assist in positioning, with supports placed beneath the patient's back and buttocks to alleviate pressure points.
  Arms: 90-degree high lateral position group
Procedure: Place the patient in the 30-degree low lateral position. — For the 30° lateral recumbent position group, patients will be rotated between left and right lateral recumbent positions at the corresponding angles every 2 hours, spending 8 hours on each side for a total treatment duration of 16 hours. During each rotation, the nursing team will ensure the patient is safely transferred from one side to the other while maintaining the prescribed lateral angle. Wedge pillows or specialized turning pads will be used to assist in positioning, with supports placed beneath the patient's back and buttocks to alleviate pressure points.
  Translated with DeepL.com (free version)
  Arms: 30-degree low lateral position group
Procedure: Place the patient in the 120-degree high lateral position. — For the 120° lateral recumbent position group, patients will be rotated between corresponding lateral recumbent positions on the left and right sides every 2 hours, spending 8 hours on each side for a total treatment duration of 16 hours. During each rotation, the nursing team will ensure the patient is safely transferred from one side to the other while maintaining the prescribed lateral angle. Wedge pillows or specialized turning pads will be used to assist in positioning, with supports placed under the patient's back and buttocks to alleviate pressure points.
  Translated with DeepL.com (free version)
  Arms: 120-degree high lateral position group
Procedure: Patients will be placed in the prone position, i.e., lying face down. — Patients will be positioned in the prone position, lying face down, with specialized prone positioning devices or pillows supporting the head and chest to ensure airway patency. Daily prone therapy duration is set according to clinical guidelines, typically lasting 16 hours.
  Arms: Prone position group

SUMMARY:
This randomized controlled trial investigates the effects of prone positioning versus lateral positioning at different angles (30°, 90°, 120°) on pulmonary function improvement in patients with acute respiratory distress syndrome (ARDS). Utilizing electrical impedance tomography (EIT) technology, the study monitors key parameters including ventilation distribution and ventilation-perfusion matching in real time, while integrating respiratory mechanics and blood gas analysis data to comprehensively evaluate the therapeutic efficacy of positional adjustments. The study hypothesizes that high-angle lateral positioning may reduce adverse complications associated with prone positioning while effectively improving oxygenation and pulmonary function. The ultimate objective is to provide a safer and more personalized positional therapy regimen for clinical practice, optimizing ARDS treatment strategies to reduce mortality and enhance patient survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. Diagnosis of ARDS according to the Berlin Definition (2023 update).
3. Clinically evaluated as suitable for positional therapy by physicians.
4. Signed informed consent obtained from the patient or legal representative.
5. Absence of severe spinal deformities or musculoskeletal disorders that may compromise safe high lateral positioning.
6. No severe skin conditions (e.g., extensive open wounds or pressure ulcers) that may affect the feasibility of lateral positioning.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Severe cardiac diseases (e.g., unstable arrhythmia or heart failure) that may worsen with positional changes.
3. Severe coagulation disorders with increased bleeding risk.
4. Known allergy to the EIT device or any of its components.
5. Severe psychiatric disorders impairing study compliance.
6. Current participation in experimental therapies that may affect pulmonary function.
7. Severe active infections requiring special isolation measures.
8. Anticipated need for emergency surgery or life-threatening complications within 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
death | One month after treatment

SECONDARY OUTCOMES:
A/P Ratio | 24 hours before treatment, 24 hours after treatment
Ventilation-Perfusion Ratio | 24 hours before treatment, 24 hours after treatment
Oxygenation index | 24 hours before treatment, 24 hours after treatment
Global Inhomogeneity Index, GI | 24 hours before treatment, 24 hours after treatment

IPD SHARING:
Plan to Share IPD: Undecided